CLINICAL TRIAL: NCT05378763
Title: A Randomized, Phase 3 Study of Poziotinib in Previously Treated Patients With Locally Advanced or Metastatic Non-Small Cell Lung Cancer (NSCLC) Harboring HER2 Exon 20 Mutations (PINNACLE)
Brief Title: A Study of Poziotinib in Previously Treated Participants With Locally Advanced or Metastatic NSCLC Harboring HER2 Exon 20 Mutations
Acronym: PINNACLE
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: The study has not enrolled any patients. The study design is under discussion and will likely be redesigned in consultation with the FDA.
Sponsor: Spectrum Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPI-POZ-301
Record Dates: First submitted 2022-05-09; First posted 2022-05-18 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: NSCLC
Keywords: Epidermal growth factor receptor (EGFR); HER2; Exon 20 mutation
MeSH Terms: interventions — HM781-36B; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Poziotinib 8 mg (Experimental): Participants will receive poziotinib 8 mg, orally, BID, in 21 day cycles or until disease progression, death, intolerable adverse events (AEs), initiation of non-protocol anti-cancer treatment, or other protocol-specified reasons for participant withdrawal from the study.
  Interventions: Drug: Poziotinib
- Docetaxel 75 mg/m^2 (Active Comparator): Participants will receive docetaxel 75 mg/m^2, intravenously (IV) on Day 1 of each 21-day treatment cycle or until disease progression, death, intolerable AEs, initiation of non-protocol anti-cancer treatment, or other protocol-specified reasons for participant withdrawal from the study.
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: Poziotinib — Poziotinib tablets
  Other Names: HM781-36
  Arms: Poziotinib 8 mg
Drug: Docetaxel — Docetaxel IV infusion
  Arms: Docetaxel 75 mg/m^2

SUMMARY:
The primary purpose of this study is to compare the progression-free survival (PFS) in participants with locally advanced or metastatic non-small cell lung cancer (NSCLC) harboring human epidermal growth factor receptor 2 (HER2) exon 20 mutations when treated with poziotinib versus docetaxel.

DETAILED DESCRIPTION:
This is a Phase 3, active-controlled, multicenter study to compare the efficacy and safety/tolerability of poziotinib versus docetaxel in previously treated participants with locally advanced or metastatic NSCLC harboring HER2 exon 20 mutations.

Participants will be randomized in a 2:1 ratio to:

* Arm A: Poziotinib 8 milligrams (mg), twice daily (BID) or
* Arm B: Docetaxel 75 milligrams per meter square (mg/m^2)

The Screening Period lasts up to 21 days prior to Cycle 1, Day 1 (C1D1). Participants will be treated in 21-day cycles or until disease progression, death, intolerable adverse events (AEs), initiation of non-protocol anti-cancer treatment, or other protocol-specified reasons.

ELIGIBILITY:
Inclusion Criteria:

Participant must:

1. Be willing and capable of providing signed and dated Informed Consent, adhering to dosing and visit schedules, and meeting the study requirements
2. Have histologically or cytologically confirmed NSCLC
3. Have at least one measurable NSCLC target lesion per RECIST v.1.1 by local assessment
4. Participant has had at least one prior systemic treatment for locally advanced or metastatic NSCLC, including platinum and a checkpoint inhibitor (CPI) therapy, unless the investigator affirms that a CPI was not medically indicated.
5. Have documentation of HER2 exon 20 mutation
6. Have an Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1
7. Have adequate hematologic, hepatic, and renal function at Baseline as per protocol

Exclusion Criteria:

Participant:

1. Has had previous treatment with poziotinib for treatment of NSCLC
2. Has EGFR or anaplastic lymphoma kinase (ALK) genome tumor alterations
3. Has had previous treatment with docetaxel for locally advanced or metastatic NSCLC. If docetaxel was received in the neo-adjuvant or adjuvant setting, progressive disease must have occurred ≥6 months after the last dose to be eligible
4. Has spinal cord compression or leptomeningeal disease
5. Has a high risk of cardiac disease, as determined by the Investigator
6. Has a history of, or signs of Grade ≥2 pneumonitis on current imaging studies
7. Is unable to take drugs orally
8. Is pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Estimated)
Dates: Start 2022-05-12 (Actual); Primary Completion 2027-12-25 (Estimated); Study Completion 2028-12-25 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Up to approximately 5 years
  PFS is defined as the time (in months) from the start of the study treatment to the date of first documented disease progression by central radiographic evaluation per the Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v.1.1) or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Overall survival (OS) | Up to approximately 5 years
  OS is defined as the time (in months) from the start of study treatment to the date of death due to any cause.
Objective Response Rate (ORR) | Up to approximately 5 years
  ORR is defined as the proportion of participants who achieve at least one complete response (CR) or partial response (PR) by the central radiographic evaluation as per the RECIST v.1.1 criteria, before disease progression. Per RECIST v.1.1 for solid tumors, CR is defined as disappearance of all tumor lesions (TLs) and disappearance or reduction of all pathological lymph nodes <10mm (short axis). PR is ≥30% decrease in sum of diameters (SOD) from Baseline.
Disease Control Rate (DCR) | Up to approximately 5 years
  DCR is defined as the proportion of participants who achieve at least one CR, PR, stable disease (SD), or non-CR/non-progressive disease (PD), by the central radiographic evaluation per the RECIST v.1.1 criteria, before disease progression. Per RECIST v.1.1 for solid tumors, CR is defined as disappearance of all tumor lesions (TLs) and disappearance or reduction of all pathological lymph nodes <10mm (short axis). PR is ≥30% decrease in sum of diameters (SOD) from Baseline, and non PD is ≥20% increase in SOD from previous smallest SOD on study, and an absolute increase of ≥5mm). SD is SOD change neither sufficient for PR nor sufficient for PD.

CONTACTS AND LOCATIONS:
Locations (1):
- Bond Clinic, P.A., Winter Haven, Florida, United States

IPD SHARING:
Plan to Share IPD: No